CLINICAL TRIAL: NCT02111551
Title: Phase I Nicotinic Agonist Treatment Trial for Autism
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: difficult to find participants and no funding
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-0614
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Autism
Keywords: Autism; Nicotinic agonist; Cognition; P50; Alpha 7
MeSH Terms: conditions — Autistic Disorder | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DMXB-A 75 mg (Experimental): DMXB-A 75 mg dose followed by a second dose of 37.5 mg at 2 hours to maintain the blood level
  Interventions: Drug: DMXB-A 150 mg; Other: placebo
- DMXB-A 150 mg (Experimental): DMXB-A 150 mg followed by a second dose of 75 mg at 2 hours to maintain the blood level
  Interventions: Other: placebo; Drug: DMXB-A 75 mg
- Sugar Pill (Placebo Comparator): placebo comparator dose followed by a second placebo dose at 2 hours to maintain blind
  Interventions: Drug: DMXB-A 150 mg; Drug: DMXB-A 75 mg

INTERVENTIONS:
Drug: DMXB-A 150 mg
  Arms: DMXB-A 75 mg; Sugar Pill
Other: placebo
  Arms: DMXB-A 150 mg; DMXB-A 75 mg
Drug: DMXB-A 75 mg
  Arms: DMXB-A 150 mg; Sugar Pill

SUMMARY:
This study plans to learn more about whether a nicotine-like investigational new drug, DMXB-A [3-(2,4-dimethoxybenzylidene) anabaseine] may have positive effects on mental focus and may help us to find new types of treatment for autism spectrum disorder. Subjects will come in for a screening visit and three more drug visits. There will be at least one week between each drug visit to allow the drug to be eliminated from your system completely. During each drug visit subjects will receive either a placebo (a capsule that looks like medicine but is not real), 75 mg of DMXB-A, or 150 mg of DMXB-A. During the drug day vital signs and well being will be monitored by the study physician. Subjects will complete some paper and pencil tasks to test memory, attention, speed, and problem solving, some rating scales and questionnaires, and the study team will record brain wave patterns with an electroencephalogram (EEG) .

ELIGIBILITY:
Inclusion Criteria:

* age 18-50
* meet DSM-5 criteria for Autism Spectrum Disorder, Levels 1 or 2, as defined by Autism Diagnostic Observation Schedule
* non-smoking persons
* in good health

Exclusion Criteria:

* persons with estimated verbal and nonverbal IQ < 70.
* abuse of other substances.
* Persons not sufficiently fluent in English to permit testing
* those with history of severe head injury
* Fragile X Syndrome
* Rett Syndrome

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference between drug and placebo on theTotal Scale Score on the repeatable Battery for the Assessment of neuropsychological Status at 2 hours after administration | 2 hours after drug administration
Difference between drug and placebo on the CPT at 30 minutes after administration | 30 minutes after drug administration
Difference between the P50 auditory evoked potential test/conditioning ratio 1 hour after administration | 1 hour after drug administration
Difference between placebo and drug on the Social Responsiveness scale 2 hours after administration | 2 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Freedman R, Olincy A, Buchanan RW, Harris JG, Gold JM, Johnson L, Allensworth D, Guzman-Bonilla A, Clement B, Ball MP, Kutnick J, Pender V, Martin LF, Stevens KE, Wagner BD, Zerbe GO, Soti F, Kem WR. Initial phase 2 trial of a nicotinic agonist in schizophrenia. Am J Psychiatry. 2008 Aug;165(8):1040-7. doi: 10.1176/appi.ajp.2008.07071135. Epub 2008 Apr 1. PMID 18381905